CLINICAL TRIAL: NCT04442334
Title: The European NAFLD Registry
Status: Recruiting | Type: Observational
Sponsor: Newcastle University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Institute of Cardiometabolism and Nutrition, France (Other); University of Cambridge (Other); Örebro University, Sweden (Other); University of Bern (Other); University of Oxford (Other); University of Turin, Italy (Other); University of Angers (Unknown); University Hospital, Antwerp (Other); Linkoeping University (Other Government); University of Helsinki (Other); UMC Utrecht (Other); National and Kapodistrian University of Athens (Other); University of Lisbon (Other); University of Milan (Other); University of Palermo (Other); Catholic University of the Sacred Heart (Other); Wuerzburg University Hospital (Other); RWTH Aachen University (Other); University of Nottingham (Other); Medical University of Vienna (Other); University of Birmingham (Other); University of Florence (Other); Assistance Publique - Hôpitaux de Paris (Other); University Medical Center Mainz (Other)
Responsible Party: Sponsor
Other Study IDs: 08759; 634413 (Other Grant/Funding Number: EU H2020); 777377 (Other Grant/Funding Number: EU H2020 IMI2)
Record Dates: First submitted 2020-05-12; First posted 2020-06-22 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: NAFLD; NASH; NASH - Nonalcoholic Steatohepatitis; Fibrosis, Liver; Steatosis of Liver; Hepatocellular Carcinoma; Cardiovascular Diseases; Type 2 Diabetes; Dyslipidaemia; Hypertension; Obesity; Other Associated Comorbidities
Keywords: NAFLD; NASH; Steatohepatitis; Liver; Cirrhosis; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Fatty Liver; Carcinoma, Hepatocellular; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Dyslipidemias; Hypertension; Obesity; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood (serum, plasma, whole blood, DNA, RNA), Liver tissue, Urine, stool, DNA, RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The LITMUS Study Cohort: Prospectively recruited NAFLD patients, recruited according to The European NAFLD Registry study protocol.
- The LITMUS Metacohort: Collated data and biological samples on patients with histologically characterised NAFLD prospectively recruited at contributing academic centres across Europe.
- EFPIA Clinical Trial Cohort: Collated data and biological samples on patients with histologically characterised NAFLD that have participated in phase 2 and phase 3 trials of IMPs for NAFLD.

SUMMARY:
The European NAFLD Registry is a prospectively recruited, observational study supporting the study of the clinical phenotype, natural history, disease outcomes and pathophysiology of Non-Alcoholic Fatty Liver Disease and Non-Alcoholic Steatohepatitis. The ultimate goals are to better understand the drivers of interpatient variation in disease pathophysiology and severity and to utilise this information to develop and validate biomarkers that, singly or in combination, enable detection and monitoring of disease progression and/or from NAFL through NASH to fibrosis and cirrhosis.

DETAILED DESCRIPTION:
The European NAFLD Registry is a major international collaboration between clinical academics at leading universities across Europe, initially established with funding from the European Association for the Study of the Liver and through the EU FP7, H2020 and IMI2 schemes to the projects FLIP (Fatty Liver Inhibition of Progression), EPoS (Elucidating Pathways of Steatohepatitis) and LITMUS (Liver Investigation: Testing marker Utility in Steatohepatitis).

The Registry is a non-interventional, observational study collecting cross-sectional and longitudinal clinical data (including clinical biochemistry/haematology, liver histology, comorbidities, prescribed medication and imaging data) and linked biological samples (Blood [Serum, Plasma], Liver Tissue, Urine, Stool) from prospectively recruited patients with NAFLD. Its purpose is to support clinical and translational research into disease pathophysiology (through development of comprehensive genetic, epigenetic, transcriptomic, metabolomic, proteomic and metagenomic datasets) and biomarker development/validation. It supports collaborative discovery science and serves as the basis for a broad international project to discover and validate biomarkers for NAFLD and associated medical conditions (LITMUS). Out-with the current study, following separate ethical approval and after separate consent, patients who have agreed to join the European NAFLD Registry may also agree to participate in a number of nested sub-studies with bi-directional sharing of data. These include the LITMUS Imaging Study, which will acquire additional imaging data across a range of modalities including, amongst others, MR-PDFF and MR-Elastography. The Registry population comprises adult patients (aged ≥18 years) with risk factors for non-alcoholic fatty liver disease (NAFLD) prospectively recruited primarily in hepatology and diabetology clinics and/or bariatric surgery units at centres across Europe. After receiving informed consent, patients will be assigned a unique study identifier (which will be used to identify all data and samples collected) which will allow all information to be recorded in a link-anonymised form.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Clinically suspected NAFLD based on any of:

   1. Patient with historical liver biopsy providing histological evidence of NAFLD or,
   2. Patient undergoing liver biopsy for suspected NAFLD with biochemical and/or radiological findings consistent with NAFLD or,
   3. Patient with radiological evidence of cirrhosis (in absence of an alternative aetiology) plus presence of ≥2 features indicative of the 'metabolic syndrome':

      * Increased waist circumference by ethnically adjusted criteria (e.g. Europid male/female ≥94cm/80cm) or overweight/obese (BMI ≥25);
      * Raised fasting glucose ≥100 mg/dL [5.6 mmol/L], HbA1c ≥48mmol/mol (6.5%) or previously diagnosed insulin resistance/type 2 diabetes mellitus (or on treatment);
      * Dyslipidaemia (fasting TG level ≥150 mg/dL [1.7 mmol/L]; or fasting HDL <40 mg/dL [1.03 mmol/L] in males and <50 mg/dL [1.29 mmol/L] in females; or on treatment);
      * Hypertension (systolic BP ≥130 or diastolic BP ≥85 mmHg, or on treatment).
3. Average alcohol consumption less than 21/14 units/week (males/females) in preceding 6 months and no history of sustained excessive consumption of alcohol in past 5 years.

Exclusion Criteria

1. Refusal or inability (lack of capacity) to give informed consent.
2. Average alcohol ingestion greater than approximately 21/14 units/week (males/females) in preceding 6 months or history of sustained excessive consumption of alcohol in past 5 years.
3. History or presence of Type 1 diabetes mellitus.
4. Presence of any other form of chronic liver disease except NAFLD.
5. Recent (within 12 months) or concomitant use of agents known to cause hepatic steatosis (long-term systemic corticosteroids [>10 days], amiodarone, methotrexate, tamoxifen, tetracycline, high dose oestrogens, valproic acid).
6. Any contra-indication to liver biopsy.
7. Recent (within 3 months) change in dose/regimen or introduction of Vitamin E (at a dose ≥400 IU/day), betaine, s-adenosyl methionine, ursodeoxycholic acid, silymarin or pentoxifylline.
8. Non-English speaking/unable to access an interpreter. Due to the nature of the study, English language or access to a relevant interpreter is a necessary criterion to ensure lifestyle (diet and exercise) and symptom data are collated.
9. Patients not meeting inclusion criteria or judged by the investigator to be unsuitable for inclusion in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a pre-existing liver biopsy providing histological evidence of NAFLD or, patients undergoing liver biopsy for suspected NAFLD with biochemical and/or radiological findings consistent with NAFLD, or patients with radiological evidence of cirrhosis (in absence of an alternative aetiology) plus presence of ≥2 features indicative of the 'metabolic syndrome'.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Detailed Characterisation of the NAFLD Patient Phenotype | 1 day
  Prospective patient recruitment and collection of cross-sectional clinical data is undertaken (including clinical biochemistry/haematology, liver histology, comorbidities, prescribed medication and imaging data).These data will be used to determine number of participants exhibiting specific features of NAFLD/NASH disease severity at enrolment including: histological grade of disease and fibrosis stage (assessed using the well validated NASH Clinical Research Network "NAFLD Activity Score" [NAS] and the FLIP "Steatosis - Activity - Fibrosis" [SAF] systems), frequency of common metabolic comorbidities (eg type 2 diabetes mellitus, dyslipidaemia, cardiovascular disease), and associated changes in clinical biochemistry/haematology/imaging parameters. Biological samples to support clinical and translational research into disease pathophysiology (e.g. genetic, epigenetic, transcriptomic, metabolomic, proteomic and metagenomic datasets) and biomarker development/validation will be collected.

SECONDARY OUTCOMES:
Disease Natural History | Through to study completion, an average of 5 years
  Longitudinal follow-up of patients with NAFLD by annual review to characterise disease natural history and determine number of participants experiencing clinically significant events including the occurrence and timing of incident comorbidities and key target conditions of interest such as:
  * Death (cause of death)
  * Major Adverse Cardiovascular Events (MACE)
  * Hepatic (e.g. diagnosis of cirrhosis, hepatic decompensation, hepatocellular carcinoma, transplantation)
  * Other (diagnosis of extra-hepatic malignancy/emergency hospitalisation)
  Routine clinical data generated as part of standard care will be collected annually. Clinical parameters assessed for changes indicative of alteration in disease state during follow-up include: clinical biochemistry/haematology, liver histology, comorbidities, prescribed medication and imaging data. Biological samples to support translational research into disease pathophysiology and biomarker development/validation will also be collected.
Lifestyle factors: Dietary Habits | Through study completion, an average of 5 years
  Cross-sectional and longitudinal study of dietary habits in patients with NAFLD using: Mediterranean Diet Score.
Lifestyle factors: Activity/Exercise | Through study completion, an average of 5 years
  Cross-sectional and longitudinal study of lifestyle factors (e.g. activity/sedentary behaviour/exercise levels) in patients with NAFLD using: International Physical Activity Questionnaire (IPAQ).
Health Related Quality of Life: CLDQ | Through study completion, an average of 5 years
  Cross-sectional and longitudinal collection of standardised data on HRQOL and symptom burden in patients with NAFLD using Patient Reported Outcome Measure (PROM): Chronic Liver Disease Questionnaire for NAFLD NASH (CLDQ NAFLD-NASH).
Health Related Quality of Life: EQ5D5L | Through study completion, an average of 5 years
  Cross-sectional and longitudinal collection of standardised data on HRQOL and symptom burden in patients with NAFLD using Patient Reported Outcome Measure (PROM): EQ-5D-5L Health
Health Related Quality of Life: NASH-CHECK | Through study completion, an average of 5 years
  Cross-sectional and longitudinal collection of standardised data on HRQOL and symptom burden in patients with NAFLD using Patient Reported Outcome Measure (PROM): NASH-CHECK.

CONTACTS AND LOCATIONS:
Overall Officials: Quentin M Anstee, MBBS, PhD, Principal Investigator — Newcastle University
Locations (37):
- Universitair Ziekenhuis Antwerpen, Antwerp, Belgium
- Helsinki University Hospital, Helsinki, Finland
- France (2):
  - Le Centre de Recherche Clinique (CRC) du CHU d'Angers, Angers
  - Institut ICAN - Institute of Cardiometabolism And Nutrition Hôpital de la Pitié Salpêtrière, Paris
- Germany (5):
  - UNIVERSITÄTSKLINIKUM der RWTH Aachen, Aachen
  - Charité University Hospital Berlin, Berlin
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg Universität Mainz, Mainz
  - Universitätsklinikums Würzburg, Würzburg
- Laiko General Hospital of Athens, Athens, Greece
- Italy (5):
  - Polytechnic University of Marche, Ancona
  - Università degli Studi Milano, Milan
  - Università di Palermo, Palermo
  - Università Cattolica del Sacro Cuore, Rome
  - Department of Medical Sciences University of Torino, Turin
- Amsterdam UMC, Amsterdam, Netherlands
- Hospital de Santa Maria, Lisbon, Portugal
- Spain (6):
  - Vall d'Hebron University Hospital, Barcelona
  - Biodonostia Health Research Institute, Donostia / San Sebastian
  - Puerta de Hierro University Hospital, Majadahonda
  - Marqués de Valdecilla University Hospital, Santander
  - Institute of Biomedicine of Sevilla (IBiS), Virgen del Rocío University Hospital, Seville
  - HU Clínico de Valladolid, Valladolid
- Sweden (2):
  - Karolinska Universitetssjukhuset, Huddinge
  - Linköping University Hospital, Linköping
- Inselspital, University Hospital, Bern, Switzerland
- United Kingdom (11):
  - University Hospitals Birmingham Nhs Foundation Trust, Birmingham
  - Addenbrooke'S Hospital, Cambridge
  - Queen Elizabeth Hospital, Gateshead
  - Hull Royal Infirmary, Hull
  - Royal London Hospital, Barts Health NHS Trust, London
  - St George's University Hospitals, London
  - The Newcastle Upon Tyne Hospitals Nhs Foundation Trust, Newcastle upon Tyne
  - Queen'S Medical Centre, Nottingham
  - Oxford University Hospitals Nhs Foundation Trust, Oxford
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGlinchey AJ, Govaere O, Geng D, Ratziu V, Allison M, Bousier J, Petta S, de Oliviera C, Bugianesi E, Schattenberg JM, Daly AK, Hyotylainen T, Anstee QM, Oresic M. Metabolic signatures across the full spectrum of non-alcoholic fatty liver disease. JHEP Rep. 2022 Mar 26;4(5):100477. doi: 10.1016/j.jhepr.2022.100477. eCollection 2022 May. PMID 35434590